CLINICAL TRIAL: NCT02884531
Title: Assessment and Treatment Responses to Patient Education and Basic Body Awareness Therapy in Hip Osteoarthritis: a Randomized Controlled Trial
Brief Title: Patient Education and Basic Body Awareness Therapy in Hip Osteoarthritis: a Randomized Controlled Trial
Acronym: HipOA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bergen (Other)
Collaborators: Haukeland University Hospital (Other); Bergen University College (Other)
Responsible Party: Principal Investigator, Liv Inger Strand, Professor, dr. philos., University of Bergen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Hip osteoarthritis RCT
Record Dates: First submitted 2016-08-22; First posted 2016-08-31 (Estimated); Last update posted 2019-10-08 (Actual); Status verified 2019-10

CONDITIONS: Hip Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Hip | interventions — Patient Education as Topic

STUDY DESIGN:
Intervention Model Description: A blinded RCT
Who Masked: Outcomes Assessor
Masking Description: The assessment at inclusion was done before randomization, and was also blinded at follow-ups
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Patient Education and BBAT (Experimental): Patients will participate in Patient Education and Basic Body Awareness Therapy
  Interventions: Other: Patient Education and Basic Body Awareness Therapy; Behavioral: Patient Education
- Patient Education (Active Comparator): Patients will only participate in Patient Education
  Interventions: Behavioral: Patient Education

INTERVENTIONS:
Other: Patient Education and Basic Body Awareness Therapy — Patient education (1/2 day) and a Physiotherapy movement modality (12 times, once a week)
  Other Names: PE and BBAT
  Arms: Patient Education and BBAT
Behavioral: Patient Education — Patient education (1/2 day)
  Other Names: PE

SUMMARY:
The incidence of hip osteoarthritis (OA) is rising in western countries due to an ageing population and the epidemic of obesity. Patients with hip OA tend to complain of hip pain and stiffness which affect alignment and mobility of the whole body and typically result in general musculoskeletal pain and disability. Clinical guidelines recommend a combination of exercise therapy, weight loss and education, adjusted to the individuals needs, to be tried out before arthroplasty eventually is offered. However, to obtain a satisfactory long-term outcome is a challenge as patients may not be motivated to comply with a training program including functional strength and mobility training, if not guided by a therapist. Basic Body Awareness Therapy (BBAT) may be an alternative training modality with a better potential for lasting effects. It is a low-impact movement therapy focusing on alignment of the body and quality of movements, implemented in daily life activities. In the BBAT learning process by doing, reflecting on and transferring body awareness into daily life movements, the investigators hypothesize that the patients will obtain self-efficacy and mastering, of importance for continued training on their own. This hypothesis will be examined in the present randomized controlled trial, comparing Patient Education combined with BBAT and Patient Education alone. The investigators will, accordingly, examine the supplementary effects of BBAT for patients with hip OA. They will also explore the importance of movement quality as observed by physiotherapist using Body Awareness Rating Scale, and how it relates to how patients perceive their movement performance. In the study the investigators will particularly address long-term effects of the intervention by comparing survival of the native hip in the two groups included in the study. Data from the study will be included in a national database of patients with non-surgical treatment of hip and knee OA (NOAR), giving rise to comparison of different movement therapies.

DETAILED DESCRIPTION:
INTRODUCTION Musculoskeletal disorders are reported to be the second largest contributor to years lived with disability worldwide, and osteoarthritis (OA) of the hips and knees among the most prevalent(1). The diagnosis of hip OA should be based on radiographic findings and symptomatic evidence (2), and a prevalence of 5.8% was reported in Norway (3). OA increases with age, every person over 60 years showing signs of osteoarthritis in at least one joint (3).

The dominant factors in OA pathogenesis is loss of articular cartilage accompanied by joint deformation, bone sclerosis, capsule shrinkage, muscle atrophy and varying degrees of synovitis (4). Physical activity is restricted by pain, and patients tend to become increasingly unfit with diminished muscle strength. Intra-articular changes are accompanied by compensatory adjustment in body posture and muscular tension, including a decrease of lumbar lordosis and thoracic kyphosis and asymmetry of the pelvis and the trunk (5). Symptoms and compensational movement adjustments have consequences for patients' daily movement and functioning, social life and self-confidence (6). A substantial increase of primary hip insertions over the last 20 years is shown in Norway by data from the Norwegian Arthroplasty Register (7). The 2014 Annual Report shows 8.099 primary hip prosthesis, and 1284 revisions, arthroplasty being more frequent in women than men (8). The risk for revisions has decreased over the years due to less aseptic loosening of prosthetic components (9), but infection is still a challenge (10).

The impact of being overweight or obese Being overweight or obese is increasingly recognized to be an important risk factor for OA in weight bearing joints (11,12). The evidence of association between obesity and development of hip OA is, however, conflicting (3,13,14). Reduction of body fat for overweight or obese people is still recommended in order to reduce both mechanical and biochemical stressors that contribute to joint degeneration (15-17).

Recommendations for non-surgical management of hip OA. There is insufficient high-quality evidence regarding non-pharmacological and nonsurgical interventions of hip OA (18-21), but clinical guidelines are rather similar in their recommendations (19,21,22).The European League Against Rheumatism (EULAR) recommends a broad range of topics like patient education, lifestyle changes, exercise modalities, weight loss, assistive technologies and adaptations, footwear and work modification, along with a biopsychosocial approach to assessment and treatment and an individualized treatment plan (21).

Patient education (PE) Empowerment of the patients by information and counseling is an important element of an up-to-date conservative treatment plan. PE was developed in Sweden by Klässbo et al. (23) aiming to empower the patients, called Better Management of Patients with Osteoarthritis (BOA www.boaregistret.se). In Sweden PE is implemented all over the country, and participation is required before total hip arthroplasty is offered (Socialstyrelsen 2012). In Denmark, PE (Good Life with osteoarthritsis in Denmark, GLA:D (www.glaid.dk ) is combined with six weeks of individualized supervised neuromuscular exercise. Even better results were shown after this program regarding pain than after BOA (24). A study examining the supplementary effects of supervised exercise vs. education alone is presently carried out on patients with severe hip OA (25). A PE called ActiveA (active living with lower limb osteoarthritis) has also been tried out for patients with hip and knee OA in Oslo (26). PE based on ActiveA principles has now been established at "Lærings- og mestringssenteret", Haukeland University Hospital (HUS) for patients with hip and knee osteoarthritis from Hordaland County.

Exercise therapy in hip OA Underlying mechanisms of beneficial effects of non-surgical treatment of hip OA are scarcely understood. Irrespective of joint, there is no evidence for effect of exercise on the pathogenesis of OA (27). It is suggested that exercise works by stabilizing the surrounding musculature of the OA-affected joint. As muscle weakness disposes to osteoarthritis, exercises may halt the progression of the disease. Endurance training can enable the patient to manage weight loss, and improve general physical functioning. Beckwée et al. (28) proposed that neuromuscular, peri-articular, intra-articular, general fitness and health, and psychosocial components might explain exercise induced improvements of pain and function.The scientific evidence for recommending therapeutic exercises for hip OA has been examined in several systematic reviews and meta-analysis (18, 29-35). Strong evidence is claimed for beneficial effects of both land- and water based aerobic and strengthening exercise programs in adults with mild to moderate OA (35), but this applies mainly to short-term effects. Some RCTs were not able to show a difference in long-term change of pain between patients who received PE combined with traditional exercises or manual therapy, versus PE alone (36, 37) or sham therapy (38). Svege et al. (39) demonstrated, however, that PE and exercises combined might postpone arthroplasty.

Recommendations are made that therapeutic exercise programs for hip or knee OA should focus on strengthening of the entire lower limb and the use of non-weight bearing exercises are questioned (32). Neuromuscular training is recommended, aiming to restore neutral functional alignment of the lower extremities, by improving dynamic motor control and functional stability (24). Although physical exercise programs are primarily recommended for patients in the early phase of OA, there is presently moderate quality evidence that preoperative exercise improves function prior to and after THA (40, 41).

How can Basic Body Awareness Therapy (BBAT) have a beneficial effect in patients with hip OA?

Empowering the patient by movement awareness learning is considered important to transform dysfunctional movements into more functional movement habits (42-44). Concrete strategies are used in BBAT to improve quality of movement in daily life. Long-lasting conditions, such as hip OA, affect multiple aspects of a persons' ability to move and function. Integrated in the BBAT program are aspects from four perspectives of human movement; biomechanical, physiological, psych-socio-cultural and existential, and movement awareness is considered a prerequisite for movement quality. Basic elements in human movement such as relating to the ground and vertical axis, freeing the breathing and finding the appropriate amount of energy required for a task, are implemented in BBAT. Movements are carried out while lying, sitting, standing, walking and also in interplay with another person (45,46). Between the Basic Body Awareness Therapy sessions, the patients are encouraged to practice movements by a) implementing the training program at home, and b) implementing quality of movements into daily life situations.

BBAT is organized as a group intervention (47, 48), and the focus is on the participants' own search for more optimal balance, core stability, free breathing and awareness, addressing movement coordination of the whole body. Evaluation of the therapy progress is done continuously by the physiotherapist together with the patients.

Pilot study A pilot study of seven patients with hip OA, taking part in Patient Education (2 hours) and Basic Body Awareness Therapy (12 times 1.5 hours weekly), was undertaken in 2014. After four months, four of seven patients demonstrated clinical significant less pain during walking. At follow-up six months later, three of five patients still reported clinical significant less pain during walking (two drop-outs unrelated to hip problem). One patient reported to be unchanged and one worse, both having minimum joint space = 0. Only the patient who reported to be worse was motivated for surgery after 10 months.

Aim for the RCT study:

To examine the supplementary effect of BBAT in patients with hip OA, by comparing the effect of Patient Education alone with Patient Education and BBAT combined.

METHOD Design The randomized controlled trial will include patients with primary hip OA randomized to one of two study arms; 1) Patient Education and Basic Body Awareness Therapy, or 2) Patient Education only.

Participants Patients with verified hip OA (by x-rays and clinical symptoms) are recruited among patients who are referred from Primary Health Care to Orthopedic department at Haukeland University Hospital to participate in Patient Education at "Lærings- og mestringssenteret". Written informed consent is a prerequisite for participation.

Sample size Pain by Numeric Rating Scale (scale 0-100): The expected difference in change between the groups is 17 points on the 0-100 Numeric Rating Scale, which is considered the minimum important difference in improvement (53). Based on a previous study (54), the investigators assume a between-participant standard deviation of change of 30 points. The required sample size, with 80% power and type I error of 0.05 is 44 in each group. Allowing for a 15% drop-out, a total of 100 patients is required.

Disability by the HOOS ADL subscale (0-100): Seventy four patients are needed to detect a clinically significant change of 10 points on the HOOS ADL subscale with SD=30, power=0.80 and alpha= 0.05 (55).100 patients will accordingly be a sufficient sample size for HOOS.

Randomization and blinding: A computer-generated block randomization schedule is used to allocate participants into one of two groups after 1) given written informed consent to participate in the study, 2) having filled in questionnaires and been tested by a blinded assessor, and 3) having participated PE. A research coordinator not involved in the randomization procedure, prepares opaque envelopes with allocation to groups.

Interventions Patient Education: The overall focus of Patient Education is empowerment of the patients by increasing their knowledge of the hip OA condition and learning how to deal with it. The patients' own experiences with hip OA and active sharing in the group will be in the forefront. Basic Body awareness Therapy (BBAT): BBAT will be implemented as a group therapy (48). A group will include 5-10 patients, be led by a specialist physiotherapist qualified in BBAT, and offered once a week. Each session last for 90 minutes, and includes movement practice (70 minutes) followed by talk (20 minutes) to let the group members share movement experiences. The participants are consecutively admitted to the class, and participate in 12 sessions. In this way experienced participants will share experiences and motivate novices. BBAT will be offered as group therapy in Primary Health Care.

Analysis of RCT: Comparison of change between the randomized groups will be performed by linear regression (ANCOVA) analysis, controlling for baseline scores. Per protocol and intention-to-treat analysis will be performed.

Ethical considerations: The project is conducted in conformity with the "Declaration of Helsinki". Approval from the Regional Ethical Committee was recived in September 2015.

ELIGIBILITY:
Inclusion Criteria:

* Women and men with primary OA according to the American College of Rheumatology Clinical Criteria, living in Bergen or within a reasonable travelling distance (judged by the patients).

Exclusion Criteria:

* Other known major physical or mental problems or disease that precludes movement training and participation in an educational program, known drug abuse, not speaking or understanding Norwegian language, pregnancy 5-9 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Numeric Rating Scale, change in pain | Baseline, 4 months and 1 year
  Pain intensity during walking
Hip disability and Osteoarthritis Outcome Score (HOOS), change in ADL | Baseline, 4 months and 1 year
  Self-reported disability

SECONDARY OUTCOMES:
Harris Hip Score (HHS) | Baseline, 4 months and 1 year
  Assesses hip disabilities and effect of treatment on four domains
The EuroQol (EQ-5D-5L) | Baseline, 4 months and 1 year
  A generic health index comprising a five-part questionnaire and a visual analogue self-rating scale
Arthritis Self-efficacy Scale (ASES) | Baseline, 4 months and 1 year
  A questionnaire about self-efficacy regarding pain and symptoms
The Patient Global Impression of Change (PGIC) | 4 months and 1 year
  Assesses the patients' own impression of change over time
6-minutes walking - test | Baseline, 4 months
  Walking distance (inside) during the time limit of 6 minutes
Chair test. | Baseline, 4 months
  The patient repeats rising up from a chair and sitting down during 30 seconds and the number is counted
Stairs test. | Baseline, 4 months
  The number of seconds used to walk up and down 18 steps x 3 is measured
Body Awareness Rating Scale (BARS) | Baseline, 4 months
  Consists of two assessment parts: 1) observation and assessment of movement quality based on 12 movements and 2) interview with the patient about movement awareness immediately after exploring each movement.
UCLA Activity Score | Baseline, 4 months and 1 year
  Assesses degree of Activity on ordinal scale

CONTACTS AND LOCATIONS:
Overall Officials: Liv I Strand, Dr.philos., Principal Investigator — University of Bergen
Locations (1):
- University of Bergen, Bergen, Norway

IPD SHARING:
Plan to Share IPD: Yes
After the RCT has been completed, the plan is to enter data in a national register for patients with osteoarthritis, NOAR. The patients give their consent to this.
Time Frame: The data will be available from January 2021 to January 2023
Access Criteria: All data that has relevance to NOAR will be shared

REFERENCES:
- [Background] Pereira D, Peleteiro B, Araujo J, Branco J, Santos RA, Ramos E. The effect of osteoarthritis definition on prevalence and incidence estimates: a systematic review. Osteoarthritis Cartilage. 2011 Nov;19(11):1270-85. doi: 10.1016/j.joca.2011.08.009. Epub 2011 Aug 24. PMID 21907813
- [Background] Grotle M, Hagen KB, Natvig B, Dahl FA, Kvien TK. Obesity and osteoarthritis in knee, hip and/or hand: an epidemiological study in the general population with 10 years follow-up. BMC Musculoskelet Disord. 2008 Oct 2;9:132. doi: 10.1186/1471-2474-9-132. PMID 18831740
- [Background] Veje K, Hyllested JL, Ostergaard K. [Osteoarthritis. Pathogenesis, clinical features and treatment]. Ugeskr Laeger. 2002 Jun 10;164(24):3173-9. Danish. PMID 12082761
- [Background] Truszczynska A, Drzal-Grabiec J, Rapala K, Tarnowski A, Gorniak K, Bialecki J. Characteristics of selected parameters of body posture in patients with hip osteoarthritis. Ortop Traumatol Rehabil. 2014 May-Jun;16(3):351-60. doi: 10.5604/15093492.1112959. PMID 25058110
- [Background] Dosanjh S, Matta JM, Bhandari M; Anterior THA Research Collaborative. The final straw: a qualitative study to explore patient decisions to undergo total hip arthroplasty. Arch Orthop Trauma Surg. 2009 Jun;129(6):719-27. doi: 10.1007/s00402-008-0671-1. Epub 2008 Jun 17. PMID 18560849
- [Background] Espehaug B, Furnes O, Engesaeter LB, Havelin LI. Hip arthroplasty in Norway 1989-2008. Tidsskr Nor Laegeforen. 2011 Aug 23;131(16):1543-8. doi: 10.4045/tidsskr.09.1091. English, Norwegian. PMID 21866193
- [Background] Fevang BT, Lie SA, Havelin LI, Engesaeter LB, Furnes O. Improved results of primary total hip replacement. Acta Orthop. 2010 Dec;81(6):649-59. doi: 10.3109/17453674.2010.537807. PMID 21110699
- [Background] Dale H, Fenstad AM, Hallan G, Havelin LI, Furnes O, Overgaard S, Pedersen AB, Karrholm J, Garellick G, Pulkkinen P, Eskelinen A, Makela K, Engesaeter LB. Increasing risk of prosthetic joint infection after total hip arthroplasty. Acta Orthop. 2012 Oct;83(5):449-58. doi: 10.3109/17453674.2012.733918. PMID 23083433
- [Background] Jiang L, Rong J, Wang Y, Hu F, Bao C, Li X, Zhao Y. The relationship between body mass index and hip osteoarthritis: a systematic review and meta-analysis. Joint Bone Spine. 2011 Mar;78(2):150-5. doi: 10.1016/j.jbspin.2010.04.011. Epub 2010 Jun 30. PMID 20580591
- [Background] Viester L, Verhagen EA, Oude Hengel KM, Koppes LL, van der Beek AJ, Bongers PM. The relation between body mass index and musculoskeletal symptoms in the working population. BMC Musculoskelet Disord. 2013 Aug 12;14:238. doi: 10.1186/1471-2474-14-238. PMID 23937768
- [Background] Apold H, Meyer HE, Espehaug B, Nordsletten L, Havelin LI, Flugsrud GB. Weight gain and the risk of total hip replacement a population-based prospective cohort study of 265,725 individuals. Osteoarthritis Cartilage. 2011 Jul;19(7):809-15. doi: 10.1016/j.joca.2011.03.013. Epub 2011 Apr 12. PMID 21524707
- [Background] Mork PJ, Holtermann A, Nilsen TI. Effect of body mass index and physical exercise on risk of knee and hip osteoarthritis: longitudinal data from the Norwegian HUNT Study. J Epidemiol Community Health. 2012 Aug;66(8):678-83. doi: 10.1136/jech-2011-200834. Epub 2012 Apr 17. PMID 22511797
- [Background] Vincent HK, Heywood K, Connelly J, Hurley RW. Obesity and weight loss in the treatment and prevention of osteoarthritis. PM R. 2012 May;4(5 Suppl):S59-67. doi: 10.1016/j.pmrj.2012.01.005. PMID 22632704
- [Background] Paans N, van den Akker-Scheek I, Dilling RG, Bos M, van der Meer K, Bulstra SK, Stevens M. Effect of exercise and weight loss in people who have hip osteoarthritis and are overweight or obese: a prospective cohort study. Phys Ther. 2013 Feb;93(2):137-46. doi: 10.2522/ptj.20110418. Epub 2012 Sep 27. PMID 23023813
- [Background] Scotece M, Conde J, Gomez R, Lopez V, Lago F, Gomez-Reino JJ, Gualillo O. Beyond fat mass: exploring the role of adipokines in rheumatic diseases. ScientificWorldJournal. 2011;11:1932-47. doi: 10.1100/2011/290142. Epub 2011 Oct 25. PMID 22194660
- [Background] Moe RH, Haavardsholm EA, Christie A, Jamtvedt G, Dahm KT, Hagen KB. Effectiveness of nonpharmacological and nonsurgical interventions for hip osteoarthritis: an umbrella review of high-quality systematic reviews. Phys Ther. 2007 Dec;87(12):1716-27. doi: 10.2522/ptj.20070042. Epub 2007 Sep 25. PMID 17906289
- [Background] Hochberg MC, Altman RD, April KT, Benkhalti M, Guyatt G, McGowan J, Towheed T, Welch V, Wells G, Tugwell P; American College of Rheumatology. American College of Rheumatology 2012 recommendations for the use of nonpharmacologic and pharmacologic therapies in osteoarthritis of the hand, hip, and knee. Arthritis Care Res (Hoboken). 2012 Apr;64(4):465-74. doi: 10.1002/acr.21596. PMID 22563589
- [Background] Roos EM, Juhl CB. Osteoarthritis 2012 year in review: rehabilitation and outcomes. Osteoarthritis Cartilage. 2012 Dec;20(12):1477-83. doi: 10.1016/j.joca.2012.08.028. Epub 2012 Sep 7. PMID 22960093
- [Background] Fernandes L, Hagen KB, Bijlsma JW, Andreassen O, Christensen P, Conaghan PG, Doherty M, Geenen R, Hammond A, Kjeken I, Lohmander LS, Lund H, Mallen CD, Nava T, Oliver S, Pavelka K, Pitsillidou I, da Silva JA, de la Torre J, Zanoli G, Vliet Vlieland TP; European League Against Rheumatism (EULAR). EULAR recommendations for the non-pharmacological core management of hip and knee osteoarthritis. Ann Rheum Dis. 2013 Jul;72(7):1125-35. doi: 10.1136/annrheumdis-2012-202745. Epub 2013 Apr 17. PMID 23595142
- [Background] Walsh NE, Brooks P, Hazes JM, Walsh RM, Dreinhofer K, Woolf AD, Akesson K, Lidgren L; Bone and Joint Decade Task Force for Standards of Care for Acute and Chronic Musculoskeletal Pain. Standards of care for acute and chronic musculoskeletal pain: the Bone and Joint Decade (2000-2010). Arch Phys Med Rehabil. 2008 Sep;89(9):1830-45. doi: 10.1016/j.apmr.2008.04.009. PMID 18760171
- [Background] Klassbo M, Larsson G, Harms-Ringdahl K. Promising outcome of a hip school for patients with hip dysfunction. Arthritis Rheum. 2003 Jun 15;49(3):321-7. doi: 10.1002/art.11110. PMID 12794786
- [Background] Skou ST, Odgaard A, Rasmussen JO, Roos EM. Group education and exercise is feasible in knee and hip osteoarthritis. Dan Med J. 2012 Dec;59(12):A4554. PMID 23290290
- [Background] Jensen C, Roos EM, Kjaersgaard-Andersen P, Overgaard S. The effect of education and supervised exercise vs. education alone on the time to total hip replacement in patients with severe hip osteoarthritis. A randomized clinical trial protocol. BMC Musculoskelet Disord. 2013 Jan 14;14:21. doi: 10.1186/1471-2474-14-21. PMID 23311889
- [Background] Svege I, Nordsletten L, Fernandes L, Risberg MA. Exercise therapy may postpone total hip replacement surgery in patients with hip osteoarthritis: a long-term follow-up of a randomised trial. Ann Rheum Dis. 2015 Jan;74(1):164-9. doi: 10.1136/annrheumdis-2013-203628. Epub 2013 Nov 19. PMID 24255546
- [Background] Pedersen BK, Saltin B. Evidence for prescribing exercise as therapy in chronic disease. Scand J Med Sci Sports. 2006 Feb;16 Suppl 1:3-63. doi: 10.1111/j.1600-0838.2006.00520.x. PMID 16451303
- [Background] Beckwee D, Vaes P, Cnudde M, Swinnen E, Bautmans I. Osteoarthritis of the knee: why does exercise work? A qualitative study of the literature. Ageing Res Rev. 2013 Jan;12(1):226-36. doi: 10.1016/j.arr.2012.09.005. Epub 2012 Sep 28. PMID 23026409
- [Background] Fransen M, McConnell S, Bell M. Exercise for osteoarthritis of the hip or knee. Cochrane Database Syst Rev. 2003;(3):CD004286. doi: 10.1002/14651858.CD004286. PMID 12918008
- [Background] McNair PJ, Simmonds MA, Boocock MG, Larmer PJ. Exercise therapy for the management of osteoarthritis of the hip joint: a systematic review. Arthritis Res Ther. 2009;11(3):R98. doi: 10.1186/ar2743. Epub 2009 Jun 25. PMID 19555502
- [Background] Fransen M, McConnell S, Hernandez-Molina G, Reichenbach S. Exercise for osteoarthritis of the hip. Cochrane Database Syst Rev. 2014 Apr 22;2014(4):CD007912. doi: 10.1002/14651858.CD007912.pub2. PMID 24756895
- [Background] Fransen M, McConnell S, Hernandez-Molina G, Reichenbach S. Does land-based exercise reduce pain and disability associated with hip osteoarthritis? A meta-analysis of randomized controlled trials. Osteoarthritis Cartilage. 2010 May;18(5):613-20. doi: 10.1016/j.joca.2010.01.003. Epub 2010 Feb 10. PMID 20188228
- [Background] Escalante Y, Saavedra JM, Garcia-Hermoso A, Silva AJ, Barbosa TM. Physical exercise and reduction of pain in adults with lower limb osteoarthritis: a systematic review. J Back Musculoskelet Rehabil. 2010;23(4):175-86. doi: 10.3233/BMR-2010-0267. PMID 21079296
- [Background] Golightly YM, Allen KD, Caine DJ. A comprehensive review of the effectiveness of different exercise programs for patients with osteoarthritis. Phys Sportsmed. 2012 Nov;40(4):52-65. doi: 10.3810/psm.2012.11.1988. PMID 23306415
- [Background] Tak E, Staats P, Van Hespen A, Hopman-Rock M. The effects of an exercise program for older adults with osteoarthritis of the hip. J Rheumatol. 2005 Jun;32(6):1106-13. PMID 15940775
- [Background] Fernandes L, Storheim K, Sandvik L, Nordsletten L, Risberg MA. Efficacy of patient education and supervised exercise vs patient education alone in patients with hip osteoarthritis: a single blind randomized clinical trial. Osteoarthritis Cartilage. 2010 Oct;18(10):1237-43. doi: 10.1016/j.joca.2010.05.015. Epub 2010 Jul 13. PMID 20633669
- [Background] Poulsen E, Hartvigsen J, Christensen HW, Roos EM, Vach W, Overgaard S. Patient education with or without manual therapy compared to a control group in patients with osteoarthritis of the hip. A proof-of-principle three-arm parallel group randomized clinical trial. Osteoarthritis Cartilage. 2013 Oct;21(10):1494-503. doi: 10.1016/j.joca.2013.06.009. Epub 2013 Jun 21. PMID 23792189
- [Background] Bennell KL, Egerton T, Martin J, Abbott JH, Metcalf B, McManus F, Sims K, Pua YH, Wrigley TV, Forbes A, Smith C, Harris A, Buchbinder R. Effect of physical therapy on pain and function in patients with hip osteoarthritis: a randomized clinical trial. JAMA. 2014 May 21;311(19):1987-97. doi: 10.1001/jama.2014.4591. PMID 24846036
- [Background] Wallis JA, Taylor NF. Pre-operative interventions (non-surgical and non-pharmacological) for patients with hip or knee osteoarthritis awaiting joint replacement surgery--a systematic review and meta-analysis. Osteoarthritis Cartilage. 2011 Dec;19(12):1381-95. doi: 10.1016/j.joca.2011.09.001. Epub 2011 Sep 10. PMID 21959097
- [Background] Gill SD, McBurney H. Does exercise reduce pain and improve physical function before hip or knee replacement surgery? A systematic review and meta-analysis of randomized controlled trials. Arch Phys Med Rehabil. 2013 Jan;94(1):164-76. doi: 10.1016/j.apmr.2012.08.211. Epub 2012 Sep 4. PMID 22960276
- [Background] Greenfield BH, Jensen GM. Understanding the lived experiences of patients: application of a phenomenological approach to ethics. Phys Ther. 2010 Aug;90(8):1185-97. doi: 10.2522/ptj.20090348. Epub 2010 Jun 10. PMID 20539020
- [Background] Jensen GM. Learning: what matters most. Phys Ther. 2011 Nov;91(11):1674-89. doi: 10.2522/ptj.2011.mcmillan.lecture. Epub 2011 Sep 8. No abstract available. PMID 21903733
- [Background] Dropsy J. Den harmoniska kroppen - en osynlig övning. Stocholm, Bokforlaget Natur och Kultur Sverige, 1983.
- [Background] Skjaerven LH, Kristoffersen K, Gard G. An eye for movement quality: a phenomenological study of movement quality reflecting a group of physiotherapists' understanding of the phenomenon. Physiother Theory Pract. 2008 Jan-Feb;24(1):13-27. doi: 10.1080/01460860701378042. PMID 18300105
- [Background] Skjaerven LH, Kristoffersen K, Gard G. How can movement quality be promoted in clinical practice? A phenomenological study of physical therapist experts. Phys Ther. 2010 Oct;90(10):1479-92. doi: 10.2522/ptj.20090059. Epub 2010 Aug 5. PMID 20688872
- [Background] Skatteboe UB, Friis S, Hope MK, Vaglum P. Body awareness group therapy for patients with personality disorders. 1. Description of the therapeutic method. Psychother Psychosom. 1989;51(1):11-7. doi: 10.1159/000288128. PMID 2602527
- [Background] Yalom I. The Theory and Practise of Group Psychotherapy. 3 ed. New York NY: Basic Books; 1995.
- [Background] Giorgi A. The theory, practice and evaluation of the phenomenological method as a qualitative research procedure. Journal of Phenomenological Psychology; 28 (2), 235-260, 1997.
- [Background] Altman R, Alarcon G, Appelrouth D, Bloch D, Borenstein D, Brandt K, Brown C, Cooke TD, Daniel W, Feldman D, et al. The American College of Rheumatology criteria for the classification and reporting of osteoarthritis of the hip. Arthritis Rheum. 1991 May;34(5):505-14. doi: 10.1002/art.1780340502. PMID 2025304
- [Background] Jensen MP, Karoly P, Braver S. The measurement of clinical pain intensity: a comparison of six methods. Pain. 1986 Oct;27(1):117-126. doi: 10.1016/0304-3959(86)90228-9. PMID 3785962
- [Background] Farrar JT, Young JP Jr, LaMoreaux L, Werth JL, Poole MR. Clinical importance of changes in chronic pain intensity measured on an 11-point numerical pain rating scale. Pain. 2001 Nov;94(2):149-158. doi: 10.1016/S0304-3959(01)00349-9. PMID 11690728
- [Background] Tubach F, Ravaud P, Baron G, Falissard B, Logeart I, Bellamy N, Bombardier C, Felson D, Hochberg M, van der Heijde D, Dougados M. Evaluation of clinically relevant changes in patient reported outcomes in knee and hip osteoarthritis: the minimal clinically important improvement. Ann Rheum Dis. 2005 Jan;64(1):29-33. doi: 10.1136/ard.2004.022905. Epub 2004 Jun 18. PMID 15208174
- [Background] Villadsen A, Overgaard S, Holsgaard-Larsen A, Christensen R, Roos EM. Immediate efficacy of neuromuscular exercise in patients with severe osteoarthritis of the hip or knee: a secondary analysis from a randomized controlled trial. J Rheumatol. 2014 Jul;41(7):1385-94. doi: 10.3899/jrheum.130642. Epub 2014 Jun 15. PMID 24931956
- [Background] Nilsdotter AK, Lohmander LS, Klassbo M, Roos EM. Hip disability and osteoarthritis outcome score (HOOS)--validity and responsiveness in total hip replacement. BMC Musculoskelet Disord. 2003 May 30;4:10. doi: 10.1186/1471-2474-4-10. Epub 2003 May 30. PMID 12777182
- [Background] EuroQol Group. EuroQol--a new facility for the measurement of health-related quality of life. Health Policy. 1990 Dec;16(3):199-208. doi: 10.1016/0168-8510(90)90421-9. PMID 10109801
- [Background] Lorig K, Chastain RL, Ung E, Shoor S, Holman HR. Development and evaluation of a scale to measure perceived self-efficacy in people with arthritis. Arthritis Rheum. 1989 Jan;32(1):37-44. doi: 10.1002/anr.1780320107. PMID 2912463
- [Background] Lauridsen HH, Hartvigsen J, Korsholm L, Grunnet-Nilsson N, Manniche C. Choice of external criteria in back pain research: Does it matter? Recommendations based on analysis of responsiveness. Pain. 2007 Sep;131(1-2):112-20. doi: 10.1016/j.pain.2006.12.023. Epub 2007 Feb 2. PMID 17276006
- [Background] Tveter AT, Dagfinrud H, Moseng T, Holm I. Health-related physical fitness measures: reference values and reference equations for use in clinical practice. Arch Phys Med Rehabil. 2014 Jul;95(7):1366-73. doi: 10.1016/j.apmr.2014.02.016. Epub 2014 Mar 5. PMID 24607837
- [Background] Skjaerven LH, Gard G, Sundal MA, Strand LI. Reliability and Validity of the Body Awareness Rating Scale (BARS), an Observational Assessment tool of Movement Quality. European Journal of Physiotherapy, 17(1), 19-21, 2015.

DOCUMENTS (1):
  • Statistical Analysis Plan (2019-09-19): https://cdn.clinicaltrials.gov/large-docs/31/NCT02884531/SAP_000.pdf